CLINICAL TRIAL: NCT01873235
Title: The Baltimore Polycystic Kidney Disease Clinical and Translational Core Study
Brief Title: PKD Clinical and Translational Core Study
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Terry Watnick, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00054815; P30DK0908; 5P30DK090868 (NIH)
Record Dates: First submitted 2013-05-23; First posted 2013-06-10 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Plasma, serum,urine, and DNA will be collected at the baseline visit and stored in a biorepository.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Main Cohort: This is an observational prospective cohort study of adults with autosomal dominant polycystic kidney disease (ADPKD) with estimated GFR at least 15cc/min/1.73m2. There are no therapeutic interventions in this observational cohort study.

SUMMARY:
Advances in our understanding of the pathogenesis of autosomal dominant polycystic kidney disease (ADPKD) have opened up possibilities of new therapies to prevent disease progression. High quality clinical investigations in patients with ADPKD, however, pose significant challenges to investigators including limited access to patients with ADPKD,insufficient guidance by experienced investigators and lack of resources to conduct these studies.

The Polycystic Kidney Disease Research Clinical and Translational Core (P30) aims to establish an infrastructure that will assist investigators in designing and conducting highest quality clinical and translational research focused on a diverse group of patients with ADPKD.

Objective 1: To establish a Mid-Atlantic cohort of ADPKD patients (N=350) with baseline clinical phenotyping performed at the General Clinical Research Unit of the University of Maryland School of Medicine.

Objective 2: To establish a state-of-the-art biobank of specimens from the ADPKD cohort including serum, plasma,urine and DNA.

Objective 3: To develop a collaborative network of physicians and practices in the Mid-Atlantic region who will contribute to the ADPKD cohort and will be willing to refer patients for future studies and trials.

Objective 4: To establish a web-based registry of ADPKD patients in the Mid-Atlantic area.

DETAILED DESCRIPTION:
The purpose of this study is to establish a prospective observational cohort of 350 well-characterized adults with ADPKD, and an associated biorepository of DNA, plasma, serum, and urine. Baseline clinical phenotyping includes measurement of renal filtration function, total kidney volume, clinical and family history, presence and history of renal and extra-renal ADPKD manifestations, cardiac function, vascular stiffness, and health-related quality of life.

Prospective characterization will include the development of ADPKD complications (e.g., infection, stones, cyst hemorrhage) and other acute medical events, and changes in symptoms and QoL.

In addition, an electronic PKD patient registry will collect demographic and contact information on adults with ADPKD interested in participating in future clinical trials and/or observational cohort studies.

No treatment interventions will be performed in these observational studies

ELIGIBILITY:
Inclusion criteria:

* Age 18 and older
* ADPKD confirmed by genetic testing or ultrasound criteria using modified Ravine criteria: with family history:several cysts per kidney (3 by sonography, 5 if by computerized tomography or MRI)without family history: 10 cysts (by any radiologic method) per kidney and exclusion of other cystic kidney diseases
* Ability to provide written informed consent prior to initiation of any study procedures and the ability in the opinion of the investigator to comply with all requirements of the study
* Glomerular Filtration Rate (GFR) greater than 15ml/min/1.73m2

Exclusion Criteria:

* End Stage Renal Disease or presently on dialysis or a prior kidney transplant

  --Pregnant, lactating, or intention to get pregnant in next 6 weeks
* Another systemic disease such as cancer or lupus
* Life expectancy less than 2 years
* Current participation in a drug treatment trial
* Non English speaking
* Uncontrolled diabetes A1C 7.0 or more within 6 months of study visit; and/or on more than one oral hypoglycemic agent
* Diabetic nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosed Polycystic Kidney Disease
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Renal volume by MRI | Baseline and 3 Year follow up measures to assess changes between the time points
  Calculations of the volume will be based on summation of the products of the area measurements of the kidneys and/or liver and slice thickness. A region-based signal threshold method will be applied to calculate total cyst volume, and the remaining parenchymal renal and hepatic volume.

SECONDARY OUTCOMES:
Quality of Life Instruments | Annually up to 3 Year follow up measures to assess changes between the time points
  Self-reported Quality of Life (pain, anxiety, depression, physical activity, fatigue).

OTHER OUTCOMES:
Hospitalizations | Annually up to 8 Year follow up to assess changes between time points
  Self- reported Hospitalizations with medical record retrieval for verification

CONTACTS AND LOCATIONS:
Overall Officials: Terry J Watnick, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine General Clinical Research Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Baltimore PKD Core Center — http://baltimorepkdcenter.org/